CLINICAL TRIAL: NCT03909724
Title: A Randomized Phase II Study of Pulsatile High-dose Sunitinib Versus TAS-102 in Patients With Metastatic Colorectal Carcinoma (mCRC)
Brief Title: Pulsatile High-dose Sunitinib Versus TAS-102 in Patients With Metastatic Colorectal Carcinoma (mCRC)
Acronym: SUNRISE-CRC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, H.M.W. Verheul, Prof. Dr. H.M.W. Verheul, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL60716.029.18.
Record Dates: First submitted 2018-12-14; First posted 2019-04-10 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Colorectal Cancer; Metastasis
Keywords: colorectal cancer; TAS-102; Sunitinib
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Sunitinib; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAS-102 (Lonsurf) (Active Comparator): 35 mg per square meter, twice daily, 5 days a week, with 2 days of rest, for 2 weeks, followed by a 14-day rest period.
  Interventions: Drug: TAS 102
- High Dose Intermittent Sunitinib (Experimental): 700 mg once every 2 weeks.
  Interventions: Drug: Sunitinib Malate

INTERVENTIONS:
Drug: Sunitinib Malate — After study inclusion, patients will be randomized (1:1) via a centralized randomization system to receive either oral sunitinib (700 mg once every 2 weeks) or TAS-102 (35 mg per square meter, twice daily, 5 days a week, with 2 days of rest, for 2 weeks, followed by a 14-day rest period). Patients will receive treatment until disease progression or discontinuation due to unacceptable toxic effects, withdrawal of consent, or other reason.
  Other Names: Sutent
  Arms: High Dose Intermittent Sunitinib
Drug: TAS 102 — After study inclusion, patients will be randomized (1:1) via a centralized randomization system to receive either oral sunitinib (700 mg once every 2 weeks) or TAS-102 (35 mg per square meter, twice daily, 5 days a week, with 2 days of rest, for 2 weeks, followed by a 14-day rest period). Patients will receive treatment until disease progression or discontinuation due to unacceptable toxic effects, withdrawal of consent, or other reason.
  Other Names: Lonsurf
  Arms: TAS-102 (Lonsurf)

SUMMARY:
The purpose of this study is to compare progression free survival rates of metastasized colorectal cancer patients refractory or intolerant to systemic therapy with fluoropyrimidine, irinotecan, oxaliplatin, anti-VEGF therapy and anti-EGFR therapy (for tumours with wild-type KRAS)); randomized for treatment with TAS-102 (standard-arm) or High Dose Intermittent Sunitinib (700 mg once every 2 weeks). The investigators hypothesis is that treatment with the experimental arm (sunitinib) will provide an improvement in progression free in this patient group.

DETAILED DESCRIPTION:
Study design: A prospective, open-label, randomized, mono-center, phase II clinical trial (with registration intent).

Hypothesis: The investigators hypothesize a clinically relevant increase in PFS by 3 months; from 2 months as reported for TAS-102 to 5 months in patients treated with sunitinib. They further hypothesize that this will result in a meaningful improvement in Quality of Life (QoL).

Primary Objective: The primary objective of this study is to improve progression free survival (PFS), of patients with metastatic colorectal carcinoma (mCRC) treated with high-dose sunitinib once every 2 weeks to 5 months, compared to the reported 2 months for TAS-102 monotherapy.

Secondary Objective: Secondary objectives include: overall survival (OS), the safety and efficacy of the treatment, the quality of life in the two study arms, the value of phosphoproteomics as a potential predictive biomarker for response to sunitinib, the potential value of blood markers for molecular diagnostics disease and response monitoring and the sensitivity, specificity.

Study Population: Patients eligible for inclusion are at least 18 years of age, with adequate organ function, who have histologically or cytologically confirmed adenocarcinoma of the colon or rectum with documented metastatic disease and have an indication for palliative treatment with TAS102 (refractory or intolerant to systemic therapy with fluoropyrimidine, irinotecan, oxaliplatin, anti-VEGF therapy and anti-EGFR therapy (for tumours with wild-type KRAS)). Major exclusion criteria include evidence of significant uncontrolled concomitant disease, previous extensive radiotherapy, recent major surgery or infection, unresolved bowel disorders and poorly controlled hypertension. All patients will provide Informed Consent prior to inclusion in the study and during the course of the trial, all relevant data will be stored in electronic Case Report Forms (eCRF).

Treatment Schedule:

After study inclusion, patients will be randomized (1:1) via a centralized randomization system to receive either oral sunitinib (700 mg once every 2 weeks) or TAS-102 (35 mg per square meter, twice daily, 5 days a week, with 2 days of rest, for 2 weeks, followed by a 14-day rest period). Patients will receive treatment until disease progression or discontinuation due to unacceptable toxic effects, withdrawal of consent, or other reason.

ELIGIBILITY:
Inclusion Criteria:

* Signed (by the patient or legally acceptable representative) and dated Informed Consent Form (ICF).
* Histological or cytological confirmed, documentation of incurable locally advanced or metastatic, colorectal adenocarcinoma, not amenable for potentially curative treatment (i.e. inoperable).
* Indication for treatment with TAS-102; progressive on (or intolerant to) therapy including fluoropyrimidine, irinotecan, oxaliplatin, anti-VEGF therapy and anti-EGFR therapy (for tumours with wild-type KRAS)).
* Evaluable disease by RECIST version 1.1 criteria (see appendix III).
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 3.
* Normal 12-lead ECG (clinically insignificant abnormalities permitted).
* No signs of clinical thyroid abnormalities (suppletion or blocking drugs permitted).
* Adequate bone marrow function
* Adequate liver function
* Albumin higher than 25 g per L
* Serum creatinine ≤1.5 x ULN
* Pregnant or breast-feeding subjects: Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. For fertile men or women of childbearing potential: documented willingness to use a highly effective means of contraception (e.g., hormonal methods [implants, injectables, or combined oral contraceptives], intrauterine devices, sexual abstinence, or vasectomized or surgically sterilized partner). Contraception is necessary for at least 6 months after receiving the study medication.

Exclusion Criteria:

* Previous treatment with sunitinib and/or TAS-102 for mCRC.
* Evidence of significant uncontrolled concomitant disease, such as cardiovascular disease (including stroke, New York Heart Association Class III or IV cardiac disease or myocardial infarction within 6 months prior to screening, unstable arrhythmia, clinically significant valvular heart disease and unstable angina); pulmonary disease (including obstructive pulmonary disease > GOLD 2 and inadequately treated symptomatic bronchospasm), and uncontrolled central nervous system, renal, hepatic, endocrine, or gastrointestinal disorders; or a serious non-healing wound or fracture.
* Extensive prior radiotherapy in the rectum, pelvis or in more than 3 vertebrae in the spine (less than 3 vertebrae are considered a small radiation field and eligibility will be decided on an individual basis from the PI).
* Poorly controlled hypertension despite adequate blood pressure medication. Blood pressure must be ≤160/95 mmHg at the time of screening on a stable antihypertensive regimen. Blood pressure must be stable on at least 2 separate measurements.
* Instable seizure disorders requiring anticonvulsant therapy.
* Major surgery, other than diagnostic surgery, within 4 weeks prior to day 1, without complete recovery.
* Uncontrolled bleeding disorders, and/or active bleeding.
* Known active bacterial, viral, fungal, mycobacterial, or other infection. (including HIV and atypical mycobacterial disease, but excluding fungal infection of the nail beds.)
* Known hypersensitivity to sunitinib, TAS-102, or to its excipients.
* Presence of any significant psychiatric disorder(s) that would interfere with the patient's compliance.
* Chemotherapy, radiotherapy, or other anti-cancer therapy within the previous 4 weeks; no nitrosoureas or mitomycin C within the previous 6 weeks; no investigational agents within the previous 4 weeks.
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis.
* Untreated or active central nervous system (CNS) metastases.
* Predisposing colonic or small bowel disorders in which the symptoms are uncontrolled as indicated by baseline of > 3 loose stools daily despite medication.
* Unresolved bowel obstruction
* Any evidence of a disease or condition that might affect compliance with the protocol or interpretation of the study results or render the patient at high risk from treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Counting from the date of study inclusion (date of randomization) to the date of progressive disease or death (1 year follow-up). Analysis after inclusion of 33% of patients (N=20)
  Counting from the date of study inclusion (date of randomization) to the date of progressive disease (or death)

SECONDARY OUTCOMES:
Overall Survival (OS) | From the date of randomization up to the date of death, assessed up to 12 months. If study medication is discontinued for any reason, survival follow-up takes place every 12 weeks, also assessed up to 12 months
  Overall Survival
Adverse events (AEs) | At the end of the study, after 12 months, the number of participants with adverse events that are related to both treatments will be assessed and compared
  Safety and tolerability of the two drugs -
Health-related quality of life (HRQoL): European Organisation for Research and Treatment of Cancer Quality of Life questionnaires (EORTC QoL) | via EORTC questionnaires, which will be filled in every 8-9 weeks (from date of randomization until the date of first documented progression or date of death, assessed up to 3 years). The questionnaires of both treatments will be assessed and compared
  European Organisation for Research and Treatment of Cancer Quality of Life questionnaires (EORTC QoL)
Liquid biopsies | The specific time points during study treatment are: (1) at baseline; (2) every 2 weeks during treatment (until progression of disease), assessed up to 12 months .
  Liquid biopsies for circulating blood biomarker analysis including microRNA and platelets containing tumor-derived RNA.

CONTACTS AND LOCATIONS:
Overall Officials: Henk Verheul, Prof. M.D., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud UMC, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Janssen JBE, Iyer KK, Gerritse SL, Janssen E, Gootjes EC, Labots M, Buffart TE, Wumkes ML, Douma JAJ, Streppel MM, Buffart LM, Jonker MA, van den Hombergh E, van Erp NP, Medema JP, Tauriello DVF, Poel D, Verheul HMW. SUNRISE-CRC: a randomized phase II study of high-dose intermittent sunitinib versus trifluridine/tipiracil in metastatic colorectal carcinoma. Oncologist. 2025 Oct 1;30(10):oyaf288. doi: 10.1093/oncolo/oyaf288. PMID 40973474